CLINICAL TRIAL: NCT03084549
Title: Study of the Analgesic Effect of the Perineal Infiltration of Ropivacaine 0.75% Versus Placebo in Post-episiotomy Perineal Pain: a Randomized, Double-blind Study
Brief Title: Study of the Analgesic Effect of the Perineal Infiltration of Ropivacaine 0.75% Versus Placebo in Post-episiotomy Perineal Pain
Acronym: ROPISIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHD065-16
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Episiotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaïne (Experimental)
  Interventions: Drug: Administration of Ropivacaïne
- Placebo (Placebo Comparator)
  Interventions: Drug: Administration of placebo

INTERVENTIONS:
Drug: Administration of Ropivacaïne — Administration of Ropivacaïne in the margins of the episiotomy
  Arms: Ropivacaïne
Drug: Administration of placebo — Administration of placebo in the margins of the episiotomy
  Arms: Placebo

SUMMARY:
Episiotomy is a common obstetric gesture (20 to 30% of deliveries by the low route). In postpartum, perineal pains associated with episiotomy are common, about 70% on D7 and persistent 13% at 5 months. Most studies of obstetrical analgesia have focussed on pain during labor or following a caesarean section. The perineal pain associated with the realization of an episiotomy has been much less studied and often undervalued.

Local ropivacaine has shown its effectiveness in the reduction of postoperative pain in many indications (wall surgery, hemorrhoidectomy, infiltration of trocar scars during laparoscopy). This product has the advantage of being well tolerated, easy access and administration. Three recent studies compared the post-episiotomy analgesic efficacy of local ropivacaine versus lidocaine versus placebo and lidocaine versus no infiltration. Two of these studies showed statistically significant results. However, they focused on the results at 24 and 48 hours and did not evaluate the analgesic efficacy in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient (≥ 18 years)
* Term ≥ 37 weeks of amenorrhea
* Right medio-lateral episiotomy performed for medical need
* Delivery of a single fetus in a cephalic presentation with or without instrumental extraction
* Delivery under epidural anesthesia
* Patient to be monitored over 6 months of study
* Patient in ability to understand protocol
* Patient having given consent and signed informed consent
* Patient with social coverage

Exclusion Criteria:

* Hypersensitivity or known allergy to Ropivacaine or to other amide-linked local anesthetics or to any of the excipients
* General contraindication specific to local anesthesia, irrespective of the local anesthetic used
* Contraindication for Ropivacaine- Obstetric paracervical anesthesia
* Hypovolemia
* Weight <50 kg
* Contra-indication or refusal of the epidural
* Poor understanding of the French language
* Substance addiction.
* Chronic pain syndrome.
* Severe hepatic or renal impairment.
* Acute porphyria.
* Caesarean section programmed.
* Tear of the 3rd degree according to the associated French classification.
* Refusal to participate in the study
* Patient under tutelage, curatorship, or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Compare the analgesic efficacy of ropivacaine 75 mg infusion versus placebo (physiological saline) in patients with right mid-lateral episiotomy during postpartum D7 delivery. | 7 days after episiotomy
  Digital pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, Principal Investigator — CHD Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Nantes, Nantes

REFERENCES:
- [Background] Cardaillac C, Ploteau S, Le Thuaut A, Dochez V, Winer N, Ducarme G. Ropivacaine 75 mg versus placebo in perineal infiltration for analgesic efficacy at mid- and long-term for episiotomy repair in postpartum women - the ROPISIO study: a two-center, randomized, double-blind, placebo-controlled trials. Trials. 2020 Jun 12;21(1):522. doi: 10.1186/s13063-020-04423-x. PMID 32532310
- [Result] Cardaillac C, Planche L, Dorion A, Ploteau S, Thubert T, Lefizelier E, Winer N, Ducarme G. Ropivacaine perineal infiltration for postpartum pain management in episiotomy repair: a double-blind, randomised, placebo-controlled trial. BJOG. 2024 Jun;131(7):899-907. doi: 10.1111/1471-0528.17266. Epub 2022 Aug 11. PMID 35876236